CLINICAL TRIAL: NCT02109640
Title: A Randomized Blinded Pilot Study to Compare Targinact vs. Oxycodone in Early Return of Gastrointestinal Function After Colorectal Surgery
Brief Title: A Comparison of Targinact vs. Oxycodone on Gut Function After Colorectal Surgery
Acronym: TACS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-005327-16
Record Dates: First submitted 2014-04-03; First posted 2014-04-10 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting
Keywords: Colorectal; Surgery; Laparoscopic; Analgesia; Enhanced Recovery; Targinact
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Agnosia | interventions — oxycodone naloxone combination; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Targinact (Experimental): Oral Targinact 10-20mg bd following laparoscopic segmental colectomy
  Interventions: Drug: Targinact; Procedure: Laparoscopic segmental colectomy
- Oxycodone (Active Comparator): Oral oxycodone 10-20mg bd following laparoscopic segmental colectomy
  Interventions: Drug: Oxycodone; Procedure: Laparoscopic segmental colectomy

INTERVENTIONS:
Drug: Targinact — Post-operative analgesia
  Other Names: Oxycodone-Naloxone
  Arms: Targinact
Drug: Oxycodone — Postoperative analgesia
  Arms: Oxycodone
Procedure: Laparoscopic segmental colectomy

SUMMARY:
Two key requirements for discharge from hospital after major abdominal surgery are adequate oral analgesia and resumption of oral nutrition. Up to 40% of patients suffer delayed discharge after abdominal surgery due to delayed return of gut function, manifesting as nausea, vomiting, constipation and abdominal distension. Opiates and their derivatives are the mainstay of postoperative analgesic regimens after abdominal surgery and are highly effective in achieving adequate pain control. However, opioids cause impaired gut function by reducing normal forward propulsion and increasing gut spasm. Opioid receptor blockers such as Alvimopan counteract these effects and can accelerate postoperative gut recovery but are expensive and cause cardiac complications; alternative painkillers such as non-steroidal anti-inflammatories are less effective than opioids and have been linked with increased risk of anastomotic leaks.

Targinact is a combination of prolonged release opioid analgesic (oxycodone hydrochloride) and naloxone hydrochloride (an opioid receptor blocker). The formulation of the product confines the naloxone action to the gut to reduce the unwanted side-effects on gut function. Targinact has been shown in patients with chronic severe pain to provide comparable analgesia to other opioid analgesics whilst reducing the unwanted side-effect of constipation.

The Investigators wish to test the hypothesis that Targinact will provide adequate analgesia after colonic resection with reduced postoperative gastrointestinal dysfunction. The surgical procedure chosen to test this hypothesis is laparoscopic segmental colectomy, a consistently reproducible intervention with a postoperative gut dysfunction rate of up to 40% (prospective data from the Edinburgh Colorectal Unit). The main outcome of the study will be return of normal gut function at the time of planned discharge (Day 3).

DETAILED DESCRIPTION:
Study hypothesis: Targinact is effective as oral analgesia after major colorectal surgery and is associated with less gut dysfunction than Oxycodone.

Up to 40% of patients suffer delayed return of gut function after elective colorectal surgery, leading to prolonged hospital stay and higher inpatient costs. For the patient, this is characterised by a variety of symptoms including nausea and vomiting, delayed ability to regain normal oral intake, abdominal discomfort/distension and constipation. Although post-operative gut dysfunction tends to resolve spontaneously in 3-7 days, both symptoms and supportive treatment (nasogastric tube insertion, repeated venous cannulation for intravenous fluid administration etc) are unpleasant.

Elective colorectal surgery is a common hospital intervention hence a reduction in the prevalence of post-operative gut dysfunction would be expected to benefit a large number of patients with attendant reduction in health service costs. The objective aligns well with the current national dissemination of Enhanced Recovery after Surgery programmes by the UK Department of Health and Scottish Government.

Post-operative gut dysfunction is multifactorial. Opioid analgesics are contributory and all Enhanced Recovery after Surgery (ERAS) programmes emphasise strategies to minimise systemic opioid use (eg using regional or local anaesthetic techniques).

Targinact has not been evaluated in the setting of short-term post operative analgesia in colorectal surgery but offers the potential to achieve effective analgesia with a lower incidence of gut dysfunction and therefore an important role within the ERAS program after colorectal surgery. Oxycodone is currently the oral opioid analgesic of choice in our unit and most patients are prescribed a combination of oxycodone and oxynorm as step-down analgesia following cessation of systemic or epidural analgesia, often in combination with fentanyl patches.

Data will be collected from patient hospital records and questionnaires administered by the principal investigator and research study nurse.

Multiple measures will be employed to record both presence of good function and absence of dysfunction.

* Time to first flatus
* Time to first bowel movement
* Time from surgery to cessation of iv fluids
* Total dose of rescue antiemetic (protocol ondansetron not included)
* Reinstitution of iv fluids (Y/N) Quantity of laxative used
* Measurement of oral nutritional intake:

Preoperative intake will be recorded by means of a recall diary. Postoperative oral intake will be recorded by the participant using a food diary for 7 days from the date of surgery. Energy intake will then be estimated using CompEat Pro® forWindows® (Nutrition Systems, Banbury, UK). Time to attain and maintain 80% of normal solid food intake and the percentage Recommended Nutritional Intake (RNI) achieved on days 1-3 and days 5-7 after surgery will be used in comparisons between study groups.

* Validated nausea and vomiting score (Miles and Wengritzky)
* Presence of abdominal distension (Y/N)
* 13C Stable Isotope Gastric Empyting Breath Test to measure gastric motility on the second postoperative morning. The technique has been previously used in the Edinburgh Department of Surgery and validated to be a reproducible and accurate measurement of upper GI motility.

Additional data to be recorded:

* Patient demographics, co morbidity, regular medications
* Pre op bowel function questionnaire
* Postoperative nausea and vomiting prediction data (Apfel score)
* Day 3 achievement of discharge criteria (pain controlled by oral analgesia, tolerating adequate oral diet and fluids, independently mobile and willing to go home) Y/N
* 30-day/Inpatient mortality
* Duration of hospital admission
* Complications (recorded by organ system and severity as assessed by Clavien/Dindo scale)
* Unscheduled readmissions to hospital within 30 days of discharge
* Patient-reported outcome questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic segmental colectomy at the Colorectal Surgery Unit, Western General Hospital, Edinburgh.

Exclusion Criteria:

* Pregnancy Age <18 years Patients lacking capacity to give informed consent. Severe liver dysfunction (Child's A or greater) Patients participating in another therapeutic clinical trial Contraindication to oxycodone, naloxone or Targinact Pre-existing dependence on opioid analgesia (current medications will be checked prior to discussing consent) Pre-existing use of opioid analgesia for chronic pain (current medications will be checked prior to discussing consent) Patients with rectal cancer Plan to form any stoma during procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh M Paterson, MD FRCS, Principal Investigator — University of Edinburgh
Locations (1):
- Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lassen K, Soop M, Nygren J, Cox PB, Hendry PO, Spies C, von Meyenfeldt MF, Fearon KC, Revhaug A, Norderval S, Ljungqvist O, Lobo DN, Dejong CH; Enhanced Recovery After Surgery (ERAS) Group. Consensus review of optimal perioperative care in colorectal surgery: Enhanced Recovery After Surgery (ERAS) Group recommendations. Arch Surg. 2009 Oct;144(10):961-9. doi: 10.1001/archsurg.2009.170. PMID 19841366
- [Background] Hendry PO, Hausel J, Nygren J, Lassen K, Dejong CH, Ljungqvist O, Fearon KC; Enhanced Recovery After Surgery Study Group. Determinants of outcome after colorectal resection within an enhanced recovery programme. Br J Surg. 2009 Feb;96(2):197-205. doi: 10.1002/bjs.6445. PMID 19160347
- [Background] Simpson K, Leyendecker P, Hopp M, Muller-Lissner S, Lowenstein O, De Andres J, Troy Ferrarons J, Bosse B, Krain B, Nichols T, Kremers W, Reimer K. Fixed-ratio combination oxycodone/naloxone compared with oxycodone alone for the relief of opioid-induced constipation in moderate-to-severe noncancer pain. Curr Med Res Opin. 2008 Dec;24(12):3503-12. doi: 10.1185/03007990802584454. PMID 19032132
- [Derived] Creamer F, Balfour A, Nimmo S, Foo I, Norrie JD, Williams LJ, Fearon KC, Paterson HM. Randomized open-label phase II study comparing oxycodone-naloxone with oxycodone in early return of gastrointestinal function after laparoscopic colorectal surgery. Br J Surg. 2017 Jan;104(1):42-51. doi: 10.1002/bjs.10322. Epub 2016 Oct 20. PMID 27762434

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 62 patients consented to study participation but 12 were not assigned to the study. This was because consent was obtained a few weeks before the date of surgery and in that interval 12 patients became ineligible (change of planned operation, presentation as emergency, development of ineligibility criteria, withdrawn from anaesthetic protocol).
Groups:
- Targinact: Oral Targinact 10-20mg bd following laparoscopic segmental colectomy
  Targinact: Post-operative analgesia
  Laparoscopic segmental colectomy
- Oxycodone: Oral oxycodone 10-20mg bd following laparoscopic segmental colectomy
  Oxycodone: Postoperative analgesia
  Laparoscopic segmental colectomy
Period: Overall Study
Arm/Group | Targinact | Oxycodone
Started | 27 | 23
Completed | 27 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Targinact | Oxycodone | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 20 | 17 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 15 | 11 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 23 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Postoperative Gut Dysfunction
Description: The proportion of participants with gut dysfunction, defined as the presence of any of the following sufficient to delay discharge on the 3rd postoperative day: nausea, vomiting, intolerance of oral intake or constipation.
Time Frame: Day 3 post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Targinact | Oxycodone
Number analyzed (Participants) | 27 | 23
Participants | 13 | 15
Statistical Analysis 1: Comparison: Targinact vs Oxycodone; Test type: Superiority or Other; p = 0.264, Fisher Exact — Absolute % difference 17.1 (95% CI -10.0,40.7); Absolute percentage difference = 17.1, 95% CI 2-sided [-10.0 to 40.7]

2. Secondary Outcome: Total Opioid Analgesia Consumption
Description: Total dose of systemic and oral Oxycodone or Targinact taken in hospital or at home until discontinued by the participant
Time Frame: Total postoperative period of analgesic consumption, an average of 1 week
Measure: Mean (Standard Deviation); unit: milligram morphine equivalents
Arm/Group | Targinact | Oxycodone
Number analyzed (Participants) | 27 | 23
milligram morphine equivalents | 78 (36) | 94 (56)
Statistical Analysis 1: Comparison: Targinact vs Oxycodone; Test type: Superiority or Other; p = 0.222, t-test, 2 sided

3. Secondary Outcome: Pain Scores
Description: Overall Benefit of Analgesia Score (OBAS): Score range 0-28 with low score=high benefit. Summed from subscales of 0-4 for the following questions:
  * Please rate your current pain at rest on a scale between 0⁄4 minimal pain and 4⁄4 maximum imaginable pain
  * Please grade any distress and bother from vomiting in the past 24 h (0⁄4 not at all to 4⁄4 very much)
  * Please grade any distress and bother from itching in the past 24 h (0⁄4 not at all to 4⁄4 very much)
  * Please grade any distress and bother from sweating in the past 24 h (0⁄4 not at all to 4⁄4 very much)
  * Please grade any distress and bother from freezing in the past 24 h (0⁄4 not at all to 4⁄4 very much)
  * Please grade any distress and bother from dizziness in the past 24 h (0⁄4 not at all to 4⁄4 very much)
  * How satisfied are you with your pain treatment during the past 24 h (0⁄4 not at all to 4⁄4 very much) Lehmann N. British Journal of Anaesthesia 105 (4): 511-18 (2010)
Time Frame: Postoperative day 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Targinact | Oxycodone
Number analyzed (Participants) | 27 | 23
units on a scale | 2 [0 to 10] | 2 [0 to 11]
Statistical Analysis 1: Comparison: Targinact vs Oxycodone; Test type: Superiority or Other; p = 0.676, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 30 days postoperative
Arm/Group | Targinact | Oxycodone
Serious Adverse Events (participants affected / at risk) | 2/27 | 0/23
Other Adverse Events (participants affected / at risk) | 19/27 | 18/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targinact (N=27) | Oxycodone (N=23)
Anastomotic leak (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intraabdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targinact (N=27) | Oxycodone (N=23)
Hypotension (Cardiac disorders) | 11 (11) | 11 (11) — Self-limiting postop
Acute urinary retention (Renal and urinary disorders) | 4 (4) | 1 (1)
Hypoxaemia postop (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Wound healing (General disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes